CLINICAL TRIAL: NCT06300671
Title: Investigation of the Effects of Different Subtalar Joint Pronation Amounts on Lower Extremity Anatomical Measurements, Jump Performances and Postural Stability in Healthy Individuals
Brief Title: The Effect of Subtalar Joint Pronation Amount on Lower Extremity Alignment and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PNSÖ-Subtalar pronation
Record Dates: First submitted 2024-02-06; First posted 2024-03-08 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Balance Disorders; Foot Injury; Lower Extremity Problem
Keywords: Subtalar joint; Hyperpronation; Kinetic Chain; Balance
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Intervention Model Description: 48 healthy individuals between the ages of 18-40 constitute the population of the study. Participants randomized into neutral, pronation, and hyperpronation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pronation Group (Active Comparator): Participants with a value between 6-9 according to the foot posture index-6 evaluation will be included in the pronation group.
  Interventions: Other: Foot Posture Index-6
- Hyperpronation Group (Active Comparator): Participants with a value between 10-12 according to the foot posture index-6 evaluation will be included in the hyperpronation group.
  Interventions: Other: Foot Posture Index-6
- Neutral Group (Active Comparator): Participants with a value between 0-5 according to the foot posture index-6 evaluation will be included in the neutral group.
  Interventions: Other: Foot Posture Index-6

INTERVENTIONS:
Other: Foot Posture Index-6 — Foot Posture Index 6 (API-6) is a clinical diagnostic tool that broadly measures whether a foot is in neutral, supination or pronation posture. During the evaluation, individuals' static standing postures in a comfortable position are observed and scored. When using API-6, researchers visually evaluate the foot according to 6 criteria, each rated on a 5-point (-2 to +2) Likert scale. Each item is scored between -2 (supination) and +2 (pronation) and 0 (for neutral position), with the total score being between -12 (high degree of supination) and +12 (high degree of pronation). The grouping of reference values showing foot posture can be summarized as follows; Neutral position from 0 to +5, pronation position from +6 to +9, hyperpronation position from +10 to +12, supination position from -1 to -5, and supination position from -6. It shows a high degree of supination position up to -12. Higher scores represent a more pronated foot posture.
  Other Names: Postural stability Assessment; Frontal Plane Projection Angle; Foot and Ankle Ability Measurement; Navicular Drop test; Weight bearing lunge test; Counter movement jump test without arm swing

SUMMARY:
The lower extremity consists of segments that can be affected by the relative position of each other. Deviation of one segment from its normal alignment in the lower extremity also affects the alignment of other segments. The hip joint can affect the frontal plane alignment from proximal to distal, while the foot and ankle complex can also affect it from distal to proximal. Increased subtalar joint pronation in the kinetic chain from distal to proximal; is associated with decreased dorsiflexion angle and increased frontal plane projection angle. It has been shown that ankle dorsiflexion limitation causes changes in the biomechanics and kinematics of landing after jumping, but no study examining the effect of foot pronation on jump tests has been found in the literature. Since the foot is located at the most distal point and acts as a support base for the kinematic chain, the smallest dynamic change in the foot affects the balance of the whole body. Due to foot pronation, changes in the sole contact surface may make it difficult for the foot to adapt to the ground, balance and postural stabilization may be adversely affected, and an increase in the workload of the muscles around the joint may be observed. In another study, it is mentioned that there is limited evidence about the effect of foot posture on postural stability. Although there are studies in the literature examining the effects of subtalar joint pronation on lower extremity alignment and postural stability, studies need to examine the effects of different subtalar joint pronation amounts on lower extremity alignment, jumping performance, and postural stability. Our study will contribute to the literature with this aspect.

DETAILED DESCRIPTION:
The foot has an important role as it supports body weight and plays a vital role during movement. The ankle complex consists of the talocrural and subtalar joints, which have diagonal axes that perform multi-planar movements. Because of its oblique axis, the subtalar joint can produce three-planar movements, pronation, and supination. Foot pronation consists of medial rotation and adduction of the talus, eversion of the calcaneus, and abduction and supination of the forefoot. Medial longitudinal arch height decreased or disappeared in feet in pronation posture. Loss of medial longitudinal arch height requires that the foot cannot absorb enough energy and must produce more force to stabilize it. In particular, abnormal alignment in the hyper pronation posture or prolonged pronation is defined as both a risk factor and an etiologic factor for increased navicular drop and malalignment patterns in the lower extremities. It is a possible etiologic cause for the development of most lower extremity overuse injuries by altering kinematics and force distribution. The lower extremity consists of segments that can be affected by the relative position of each other. Deviation of one segment from its normal alignment in the lower extremity also affects the alignment of other segments. In the frontal plane alignment, the hip joint can be affected from proximal to distal, while the foot and ankle complex can be affected from distal to proximal. Increased subtalar joint pronation in the kinetic chain from distal to proximal is associated with decreased dorsiflexion angle and increased frontal plane projection angle. It has been shown that ankle dorsiflexion limitation causes changes in the biomechanics and kinematics of landing after jumping, but no study examining the effect of foot pronation on jump tests has been found in the literature.

Since the foot is located at the most distal point and acts as a support base for the kinematic chain, the smallest dynamic change in the foot affects the balance of the whole body. Due to foot pronation, changes in the sole contact surface may make it difficult for the foot to adapt to the ground, balance and postural stabilization may be adversely affected, and an increase in the workload of the muscles around the joint may be observed. It is mentioned that there is limited evidence about the effect of foot posture on postural stability. there is a need for studies examining the effects of different subtalar joint pronation amounts on lower extremity alignment, jumping performance, and postural stability. Our study will contribute to the literature with this aspect.

ELIGIBILITY:
Inclusion Criteria:

- Being between the ages of 18-40

* Pain, difficulty in walking and loss of function, etc. not having complaints
* Foot posture index value should be between 6-12
* Not having any orthopedic disease
* Not having visual or hearing impairment
* Not having been involved in any physical therapy program in the last 6 months.
* Not having undergone any surgical procedure on the lower extremity
* Not using analgesic medication within the specified treatment days throughout the research period.

Exclusion Criteria:

* Having a lower extremity congenital anomaly
* Having a history of lower extremity surgery or planned lower extremity surgery within the next 12 months
* Having any signs of pain in the lower extremities
* Having ligament hyperlaxity
* Having a history of tendon or cartilage injury
* Having serious illnesses
* Predominant knee pain from other knee structures, hip or lumbar spine
* Having a history of using any shoe insert-orthosis-insoles or knee injection in the last 3 months
* Having any neurological or systemic inflammatory arthritis disorder (neurological involvement that affects movement)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Baseline
  Static and dynamic balance assessments The Biodex Balance System (BDS) (Biodex Medical Systems Inc., Shirley, New York, USA) will be used. Measurements will be made with bare feet. Each test will last 20 seconds and will be made in 3 measurements with 10-second rest periods. During the measurement, individuals will be asked to stand on their weight-bearing knees in 15° flexion, their non-weight-bearing contralateral knees in 90° flexion, and to look forward by crossing their arms at chest level. In dynamic balance evaluation, the difficulty level of the test will be set to 4.

SECONDARY OUTCOMES:
Frontal Plane Projection Angle | Baseline
  During the frontal plane projection angle (FPPA) measurement, a straight line will be drawn from the anterior superior spina iliaca along the femur to the midpoint of the patella, and the midpoint of the ankle will be determined as the reference point by a straight line drawn from the midpoint of the patella. Participants will stand with their feet aligned in the sagittal plane and their arms crossed across their chests. By prior instruction, subjects will be asked to squat up to 60º knee flexion in a controlled manner without losing their balance, before returning to the starting position. Digital recordings of the frontal plane will be made while individuals perform a single-leg squat test at 60º knee flexion 3 times. The FPPA degree is measured from the medial aspect of the knee and calculated by subtracting 360. FPPA of 195° and above will be considered pathological.
Foot and Ankle Ability Measurement | Baseline
  The Foot and Ankle Ability measurement scale consists of daily living activities and sports subheadings. The scale includes 29 items scored between 0 and 4. Standardized answer options are answered using five-point Likert options ranging from 0 (I cannot do it) to 4 (No difficulty). From the participants; They are asked to mark the activity as no difficulty (4 points), mild difficulty (3 points), moderate difficulty (2 points), extreme difficulty (1 point), cannot do (0 points) or N/A (not applicable). High scores; It shows more functional ability.
Navicular Drop Test | Baseline
  The navicular drop test (NDT) is a clinical method for assessing the mobility of the medial longitudinal arch (MLA). The extent of navicular subsidence is assessed to determine the flexibility of the MLA and the position of the navicular with and without transfer of body weight. To assess navicular drop, the subtalar joint will be positioned in neutral position and the height of the navicular will be measured in non-weight bearing position. Then the measurement will be repeated in weightbearing position. The height difference between the two measurements in sitting and standing is recorded as the NDT value. Values more than 10mm is accepted as pathological.
Weight bearing lunge test | Baseline
  Weight-bearing lunge test (WBLT) is frequently used in individuals with ankle instability in order to determine dorsiflexion normal joint movement. During WBLT the participant puts their hands on the wall and takes one leg forward and the other leg helps balance behind. The maximum distance that the knee touches the wall is recorded without allowing the heel of the front foot to lose contact with the ground.
Countermovement jump test without arm swing | Baseline
  In the starting position of the test, participants stood in the middle of the Optojump device with their feet hip-width apart. With hands on hips, participants were asked to squat until their thighs were parallel to the ground and then immediately jump up. Bending the hips and knees before landing; Participants were instructed to keep their hands on their hips and legs in extension, maintaining this position during the jump and even when they landed, as this would increase flight time and reduce the accuracy and reliability of the results. During testing, all participants wore sneakers. The test was repeated 3 times and the best value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PT, PhD, Principal Investigator — Bahcesehir University, Faculty of Health Sciences; Ozlem Feyzioğlu, PT, PhD, Study Chair — Acibadem Mehmet Ali Aydinlar University, Faculty of Health Sciences; Nurefşan Kaygaz, PT, Study Chair — Bahcesehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation; Yahya Süleyman Mollaibrahimoğlu, PT, Study Chair — Bahcesehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation
Locations (1):
- Bahcesehir University, Beşiktaş, Istanbul, Turkey (Türkiye)